CLINICAL TRIAL: NCT05915897
Title: Whole Blood Biospecimen Collection for Subjects With Chronic Granulomatous Disease (CGD)
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit subjects due to disease rarity
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-09687
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Chronic Granulomatous Disease
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CGD with p47phox phenotype
  Interventions: Diagnostic Test: Specimen Donation
- X-Linked CGD
  Interventions: Diagnostic Test: Specimen Donation

INTERVENTIONS:
Diagnostic Test: Specimen Donation — blood donation

SUMMARY:
The primary study objective is to collect biospecimen samples (e.g., blood) from participants diagnosed with Chronic Granulomatous Disease (CGD). The biospecimens will be used to create a biorepository that can be used to identify disease associated biomarkers and potential targets with immune and multi-omics profiling. The disease sample collection and analysis will be the foundation for an extensive network of biospecimen access and linked datasets for future translational research.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to provide written informed consent
* The participant is willing and able to provide appropriate photo identification
* Participants aged 18 to 85
* Participants have been diagnosed with Chronic Granulomatous Disease (CGD)
* Subjects who have a confirmed p47phox CGD mutation or Subjects who have a confirmed X-linked CGD mutation

Exclusion Criteria:

* Participants who are pregnant or are nursing
* Participants with a known history of HIV, hepatitis, or other infectious diseases
* Participants who have taken an investigational product in the last 30 days
* Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have been diagnosed with Chronic Granulomatous Disease (CGD)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Participants have been diagnosed with Chronic Granulomatous Disease (CGD) | 1 Year
  Participants have been diagnosed with Chronic Granulomatous Disease (CGD)

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine BioSciences, Inc., Woburn, Massachusetts, United States